CLINICAL TRIAL: NCT01213108
Title: Effects of the Örebro Prevention Program on Youth Drinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish National Institute of Public Health (Unknown); Alcohol Research Council of the Swedish Alcohol Retailing Monopoly (Unknown)
Responsible Party: Håkan Leifman, Head of Office, PhD, STAD-CPF
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HFÅ 2007/44
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Youth Drinking
Keywords: Örebro prevention program; Youth drinking
MeSH Terms: conditions — Underage Drinking | interventions — Commerce

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Örebro prevention program (Experimental)
  Interventions: Behavioral: Örebro prevention program
- Control (Active Comparator): Business as usual
  Interventions: Behavioral: Business as usual

INTERVENTIONS:
Behavioral: Örebro prevention program — 6 presentations on alcohol-specific parenting practices to parents of 13-16 year olds youth
  Arms: Örebro prevention program
Behavioral: Business as usual — Regular alcohol prevention activities and curricula in Swedish schools
  Arms: Control

SUMMARY:
The Örebro prevention program is a brief (6 x 30 minutes)program administered to parents of 13-16 year old youths in regular parental meetings. The program aims to encourage parents to maintain a restrictive attitude towards youth drinking throughout their children's teenage years, and thereby postpone and reduce youth drinking. A previous quasi-experimental study by the program developers showed a sustained alcohol-specific restrictivity among parents exposed to the program, and also a reduction on drinking measures among the youths of the exposed parents (Koutakis, Stattin & Kerr, 2008). This study aims to investigate whether these effects are sustained also when the program has gone into wide dissemination in Sweden.

ELIGIBILITY:
Inclusion Criteria: Municipal schools in counties with local ÖPP program presenters, comprising grades 7-9, with at least two 7th grade classes in parallel, and with no previous experience of the Örebro prevention program.

-

Exclusion Criteria:

-

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1752 (Actual)
Dates: Start 2007-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Self-reported drunkenness | 12 months
  Self-reported drunkenness among youth
Self-reported drunkenness | 30 months
  Self-reported drunkenness among youth

SECONDARY OUTCOMES:
Self-reported alcohol consumption | 12 months
  Self-reported alcohol consumption among youth
Self-reported alcohol consumption | 30 months
  Self-reported alcohol consumption among youth

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Bodin, PhD, Principal Investigator — Centre for Psychiatry Research Stockholm, Karolinska Institutet/Stockholm County Council Health Care Provision
Locations (1):
- STAD, Centre for Psychiatry Research Stockholm, Karolinska Institutet/Stockholm County Council Health Care Provision, Stockholm, Sweden

REFERENCES:
- [Derived] Bodin MC, Strandberg AK. The Orebro prevention programme revisited: a cluster-randomized effectiveness trial of programme effects on youth drinking. Addiction. 2011 Dec;106(12):2134-43. doi: 10.1111/j.1360-0443.2011.03540.x. Epub 2011 Sep 21. PMID 21676046